CLINICAL TRIAL: NCT03406546
Title: Comparison of Sedation and General Anesthesia With Laryngeal Mask in Therapeutic Bronchoscopy
Brief Title: Sedation Strategies for Therapeutic Bronchoscopy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The sample size should be re-calculated based on the first 20 cases.
Sponsor: Changhai Hospital (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); Ruijin Hospital (Other); Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Jia-feng Wang, MD, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SED-TFB
Record Dates: First submitted 2017-12-13; First posted 2018-01-23 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Bronchoscopy; Sedation
MeSH Terms: interventions — Dexmedetomidine; Remifentanil; Laryngeal Masks

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group DR (Experimental): Patients sedated with dexmedetomidine and remifentanil.
  Interventions: Drug: Dexmedetomidine; Drug: Remifentanil
- Group LMA (Experimental): General anesthesia was applied using laryngeal mask.
  Interventions: Device: Laryngeal mask

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine was used as a sedation agent with less side effect on respiratory system.
  Arms: Group DR
Drug: Remifentanil — Remifentanil was used to prevent cough induced by bronchoscopy.
  Arms: Group DR
Device: Laryngeal mask — Laryngeal mask was used to ensure respiration function during general anesthesia.
  Arms: Group LMA

SUMMARY:
Therapeutic bronchoscopy is a common procedure to treat respiratory diseases. The procedure includes stent implantation, bronchus dilation, electronic incision, laser therapy, and so on. Most of these procedures are painful and require general anesthesia. Conventionally, the general anesthesia for therapeutic bronchoscopy was performed using laryngeal mask. But in the previous experiences, the investigators found that sedation with dexmedetomidine and remifentanil was as effect as laryngeal mask anesthesia. The present study was performed to compare the two approach for sedation or anesthesia in therapeutic bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for flexible therapeutic bronchoscopy
* Adult patients aged 18 to 65 years
* American Society of Anesthesiologists (ASA) Physical Status Classification I-II
* BMI 18.5-25kg/m2
* Subjects provide informed consent

Exclusion Criteria:

* Severe airway obstruction
* Coagulation disorder
* Repeat bronchoscopy (more than 3 times)
* Severe liver and renal dysfunction
* Cardiovascular and cerebrovascular diseases
* Pregnancy
* Chronic opioid user
* Drug abusers or addicts

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Recovery time | After termination of the sedation medication, assessed up to 3 hours
  Duration of the recovery from sedation

SECONDARY OUTCOMES:
Satisfaction score of the patients and bronchoscopists | Across the procedure, assessed up to 3 hours
  Satisfaction score of the patients and bronchoscopists regarding to the sedation quality measured by a 0-100 visual analogue scale (VAS). 100 refers to the highest satisfaction degree while 0 refers to the worst satisfaction degree.
Prevalence of the side effects of respiratory and circulatory system | Across the sedation or anesthesia, assessed up to 3 hours
  The number of the side effects in respiratory and circulatory system during the procedure, including hypertension, hypotension, tackycardia, bradycardia, hypoxia and larynx spasm.
Cost of anesthesia or sedation | Across the sedation or anesthesia, assessed up to 3 hours
Cough score | From the completion of local anesthesia with lidocaine to the completion of bronchoscopy procedure, assessed up to 3 hours
  Cough score across the procedure will be classified into 4 degree (1-4) as follows. 1 = none, 2 = one gag or cough only, 3 = >1 gag or cough, but acceptable conditions, 4 = unacceptable conditions
The numbers of the times of body movement | From the completion of local anesthesia with lidocaine to the completion of bronchoscopy procedure, assessed up to 3 hours
  The numbers of the times of any body movement across the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Anesthesiology, Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided